CLINICAL TRIAL: NCT00644410
Title: A Single Centre, Randomised Controlled Study of the Effect of NOGA-guided Direct Intramyocardial Injection of Mesenchymal Stromal Cells on the Development of New Myocardium and Blood Vessels in Patients With Heart Failure
Brief Title: Autologous Mesenchymal Stromal Cell Therapy in Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JKastrup, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC heart failure
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Congestive Heart Failure
Keywords: heart failure; stem cell; mesenchymal stromal cell; mesenchymal stem cell
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The number of mesenchymal stromal cells reached after two culture expansion passages.
  Interventions: Biological: Mesenchymal stromal cell
- 2 (Placebo Comparator): Saline
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Mesenchymal stromal cell — Mesenchymal stromal cells 20 - 40 mill.
  Arms: 1
Biological: Saline — 12 injection with 0.2 ml saline
  Arms: 2

SUMMARY:
It is a single centre, randomised controlled study of the effect of NOGA-guided direct intramyocardial injection of mesenchymal stromal cells on the development of new myocardium and blood vessels in patients with heart failure.

Stem cells will be obtained from the bone marrow and culture expanded for 6 - 8 weeks before injected into the myocardium.

The patients will be followed with safety, clinical, MRI and CT endpoints for 1 year.

DETAILED DESCRIPTION:
The primary objective is to investigate the regenerative capacity of direct intra-myocardial injection of mesenchymal stromal cells in patients with reduced left ventricular EF (≤45%) and heart failure NYHA 2-3.

A total of 60 patients with will be enrolled in the study and randomised 2: 1 to cells or placebo (saline).

The patients will be followed for 12 months. The primary endpoint is changes in left ventricle end-systolic volume (LVESV) at 6 months follow-up.

The secondary endpoints are changes in left ventricular ejection fraction (LVEF), end-diastolic volume and end-systolic mass at 6 months follow-up.

Other secondary endpoints are NYHA, CCS, Kansas City Cardiomyopathy Questionnaire (KCCQ), 6 min walking test, and major adverse events endpoints: all-causes death, cardiovascular death, and hospitalization for worsening heart failure and MI at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* EF < 45 %
* NYHA 2 - 3

Exclusion Criteria:

* Acute coronary syndrome within last 6 weeks.
* Pregnancy
* FEV1 <1.0
* Cancer
* Any severe disease which could interfere with the treatment or the outcome

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Improvements in left ventricular function | 6 and 12 months

SECONDARY OUTCOMES:
Clinical improvements | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- The Heart Centre, Rigshospitalet University Hospital Copenhagen,, Copenhagen, Denmark

REFERENCES:
- [Derived] Mathiasen AB, Qayyum AA, Jorgensen E, Helqvist S, Fischer-Nielsen A, Kofoed KF, Haack-Sorensen M, Ekblond A, Kastrup J. Bone marrow-derived mesenchymal stromal cell treatment in patients with severe ischaemic heart failure: a randomized placebo-controlled trial (MSC-HF trial). Eur Heart J. 2015 Jul 14;36(27):1744-53. doi: 10.1093/eurheartj/ehv136. Epub 2015 Apr 29. PMID 25926562
- [Derived] Mathiasen AB, Jorgensen E, Qayyum AA, Haack-Sorensen M, Ekblond A, Kastrup J. Rationale and design of the first randomized, double-blind, placebo-controlled trial of intramyocardial injection of autologous bone-marrow derived Mesenchymal Stromal Cells in chronic ischemic Heart Failure (MSC-HF Trial). Am Heart J. 2012 Sep;164(3):285-91. doi: 10.1016/j.ahj.2012.05.026. PMID 22980293